CLINICAL TRIAL: NCT02188485
Title: Social Connections and Late Life Suicide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kimberly Van Orden, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH096936 (NIH); K23MH096936 (NIH)
Record Dates: First submitted 2014-07-02; First posted 2014-07-11 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Depression; Suicidal Ideation
MeSH Terms: conditions — Depression; Suicidal Ideation | interventions — engage 8200

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ENGAGE: a social engagement intervention (Experimental): ENGAGE is a brief psychotherapy that specifically targets increased social engagement and activity. The study will use the ENGAGE manual developed by Drs. Alexopoulos, Arean and their colleagues, focusing on increased engagement in activities that allow subjects to be social (targeting thwarted belongingness) or contribute to the well-being of others (targeting perceived burdensomeness).
  Interventions: Behavioral: ENGAGE
- Care-as-Usual (No Intervention): Care as usual in primary care with study assessments.

INTERVENTIONS:
Behavioral: ENGAGE — Up to 10 sessions delivered in the home.
  Arms: ENGAGE: a social engagement intervention

SUMMARY:
With the long-term goal of improving interventions for late-life suicide, the purpose of this study is to examine whether a mechanism by which behavioral interventions reduce risk for late-life suicide is by increasing social connectedness. The investigators propose to examine whether a manualized intervention that targets connectedness--ENGAGE--increases connectedness in older adults who report clinically significant depression and disconnectedness-operationalized as feeling lonely and/or like a burden on others. The investigators propose a randomized controlled trial comparing the ENGAGE intervention with care-as-usual (CAU), using n=100 primary care patients aged ≥ 60 years who report social disconnectedness (i.e., loneliness or burdensomeness) and either Minor or Major Depression. At baseline, 3-week, 6-week and 10-week assessments, subjects will report on social connectedness, depression, and suicide risk. The investigators hypothesize that those subjects assigned to ENGAGE will report greater increases in connectedness-measured as greater belongingness and lower burdensomeness-compared to CAU; that ENGAGE will produce greater reductions in depression and suicide ideation than CAU; and that changes in depression will be accounted for changes in social connectedness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 yrs;
* English speaking;
* Reside in the community;
* Endorse social disconnectedness, as measured by feeling lonely and/or like a burden on others;
* Meet criteria for Minor or Major Depression.

Exclusion Criteria:

* Imminent risk for suicide;
* Active psychosis;
* Significantly impaired cognitive functioning (i.e., MOCA <23);
* Active substance abuse in the last year (AUDIT score of 5 or more);
* Hearing loss that precludes comfortable communication;
* Residence in a long-term care facility.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly A Van Orden, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Result] Van Orden, K. A., et al.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from primary care and an outpatient geriatric psychiatry clinic.
Pre-assignment Details: Eligibility criteria were assessed at a baseline interview prior to randomization.
Period: Overall Study
Arm/Group | ENGAGE: a Social Engagement Intervention | Care-as-Usual
Started (Randomization) | 32 | 30
Completed | 30 | 27
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 1
Not completed — PI withdrew, lack of capacity | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ENGAGE: a Social Engagement Intervention | Care-as-Usual | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.78 (9.27) | 71.46 (8.96) | 72 (9.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 42
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 32 | 30 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 31 | 26 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 30 | 62
Depression Symptom Severity [Mean (Standard Deviation); unit: units on a scale] — Depression severity was measured with the 16-item Quick Inventory of Depressive Symptomatology (QIDS), interviewer rated version, with scores ranging from 0 to 27, with higher scores indicating greater depression (worse outcomes).
  units on a scale | 8.41 (4.32) | 7.37 (5.26) | 7.90 (4.79)
Low Belonging (INQ-TB) [Mean (Standard Deviation); unit: units on a scale] — Thwarted (low) belonging was measured by the Interpersonal Needs Questionnaire, thwarted belonging subscale (INQ-TB). Scores on the thwarted belonging subscale range from 0-18, with greater scores indicating greater thwarted belonging (i.e., worse outcome).
  units on a scale | 6.47 (3.69) | 5.97 (4.11) | 6.23 (3.87)
Perceived burden (INQ-PB) [Mean (Standard Deviation); unit: units on a scale] — Perceived burdensomeness was measured by the Interpersonal Needs Questionnaire Perceived Burden subscale (INQ-PB). Scores on the perceived burden subscale range from 0-12, with greater scores indicating greater perceived burden on others (i.e., worse outcome).
  units on a scale | 1.25 (1.98) | 1.23 (1.98) | 1.25 (1.98)
Suicide Ideation (GSIS) [Mean (Standard Deviation); unit: units on a scale] — Suicide ideation was measured by the Geriatric Suicide ideation scale, with scores ranging from 4 to 20, with greater scores indicating greater suicide ideation (i.e., worse outcome).
  units on a scale | 7.81 (3.27) | 7.77 (3.14) | 7.79 (3.18)

OUTCOME MEASURES:

1. Primary Outcome: Social Connectedness
Description: Severity of social disconnectedness at 10 weeks, operationalized as thwarted belongingness and perceived burdensomeness, measured by the Interpersonal Needs Questionnaire. Scores on the thwarted belonging subscale range from 0-18, with greater scores indicating greater thwarted belonging (i.e., worse outcome). Scores on the perceived burden subscale range from 0-12, with greater scores indicating greater perceived burden on others (i.e., worse outcome).
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | ENGAGE: a Social Engagement Intervention | Care-as-Usual
Number analyzed (Participants) | 30 | 27
score on scale
  Thwarted Belonging (INQ) | 4.33 (3.49) | 4.30 (4.30)
  Perceived burden (INQ | 0.77 (1.92) | 0.82 (1.80)
Statistical Analysis 1: Comparison: ENGAGE: a Social Engagement Intervention vs Care-as-Usual; Thwarted belonging (INQ-TB) at 10 week follow-up; Test type: Superiority; p = .278, Mixed Models Analysis; Mean Difference (Final Values) = -.79, Standard Error of Mean .72 — This mean difference is not identical to the mean difference presented in the summary table because this mean difference was adjusted for random effects in the model
Statistical Analysis 2: Comparison: ENGAGE: a Social Engagement Intervention vs Care-as-Usual; Perceived burden (INQ-PB) at 10-week follow-up; Test type: Superiority; p = .591, Mixed Models Analysis; Mean Difference (Final Values) = -.20, Standard Error of Mean .38 — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Suicide Ideation
Description: Suicide ideation at 10 weeks, measured by the Geriatric Suicide ideation scale, with scores ranging from 4 to 20, with greater scores indicating greater suicide ideation (i.e., worse outcome).
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ENGAGE: a Social Engagement Intervention | Care-as-Usual
Number analyzed (Participants) | 30 | 27
score on a scale | 6.6 (2.93) | 6.56 (3.36)
Statistical Analysis 1: Comparison: ENGAGE: a Social Engagement Intervention vs Care-as-Usual; Test type: Superiority; p = .511, Mixed Models Analysis; Mean Difference (Final Values) = -.34, Standard Error of Mean .52 — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Depression
Description: Depression severity was measured with the Quick Inventory of Depressive Symptomatology (QIDS), interviewer rated version, with scores ranging from 0 to 27, with higher scores indicating greater depression (worse outcomes).
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ENGAGE: a Social Engagement Intervention | Care-as-Usual
Number analyzed (Participants) | 30 | 27
score on a scale | 5.37 (3.63) | 6.15 (4.81)
Statistical Analysis 1: Comparison: ENGAGE: a Social Engagement Intervention vs Care-as-Usual; Test type: Superiority; p = .014, Mixed Models Analysis; Mean Difference (Final Values) = -2.47, Standard Error of Mean .85 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Participant engagement in the study (i.e., 10 weeks)
Arm/Group | ENGAGE: a Social Engagement Intervention | Care-as-Usual
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/32 | 2/30
Other Adverse Events (participants affected / at risk) | 0/32 | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENGAGE: a Social Engagement Intervention (N=32) | Care-as-Usual (N=30)
Psychiatric hospitalization (Psychiatric disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
The primary limitation was the sample size that was underpowered to detect small changes in target mechanisms and suicide ideation. A lack of assessment of social engagement in both groups limited our ability to fully examine this potential target mechanism. Aspects of the study design that increase generalizability to the population of interest also created a heterogenous sample with regards to functioning and contributors to disconnection that may reduce precision for detecting effects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-19): https://cdn.clinicaltrials.gov/large-docs/85/NCT02188485/Prot_SAP_000.pdf